CLINICAL TRIAL: NCT04356352
Title: A Comparison of Lidocaine, Esmolol, and Placebo Without Use of a Tourniquet for Relieving Pain From Intravenous Administration of Propofol
Brief Title: Lidocaine, Esmolol, or Placebo to Relieve IV Propofol Pain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: feasibility of enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00063576
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Injection Site Irritation; Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; esmolol

STUDY DESIGN:
Intervention Model Description: subjects randomized to receive either lidocaine, esmolol, or placebo immediately prior to the administration of propofol for their surgical procedure to treat injection site pain caused by propofol
Who Masked: Participant, Care Provider
Masking Description: assessor asking for pain scores will be blinded from the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine (Active Comparator): 1 mg/kg lidocaine to a max of 100 mg
  Interventions: Drug: Lidocaine
- Esmolol (Active Comparator): 0.5 mg/kg esmolol to a max of 50 mg
  Interventions: Drug: Esmolol
- Placebo (Placebo Comparator): Saline water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine — 1 mg/kg lidocaine to a max of 100 mg administered approximately 30 seconds prior to the administration of propofol, with pain score obtained before the propofol is administered.
  Arms: Lidocaine
Drug: Esmolol — 0.5 mg/kg esmolol to a max of 50mg administered approximately 30 seconds prior to the administration of propofol, with pain score obtained before the propofol is administered.
  Arms: Esmolol
Other: Placebo — saline water administered approximately 30 seconds prior to the administration of propofol, with pain score obtained before the propofol is administered.
  Arms: Placebo

SUMMARY:
The primary hypothesis is that esmolol and lidocaine, when given without the use of a tourniquet, provide relief of propofol injection pain that is superior to placebo when assessed using the propofol pain scoring tool

DETAILED DESCRIPTION:
The study will include three arms: lidocaine, esmolol, and placebo. Eligible patients will be 18-60 years old, ASA physical status 1-3, and scheduled for an elective surgical procedure. Patients will be randomized to receive lidocaine, esmolol, or placebo. Both the patients and the administering/observing providers will be blinded to the study drug or placebo being administered

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* ASA 1-3
* Elective surgical procedure

Exclusion Criteria:

* BMI ≥ 45
* Pregnancy
* Requirement for RSI or awake intubation
* Suspected or known difficult airway
* Contraindication to IV in either upper extremity
* Chronic pain syndrome including fibromyalgia
* Use of opioids, NSAIDs, or other analgesics within 24 hours (including preoperative PO Celebrex, Lyrica, Tylenol, etc.)
* Any use of opioids in the past three months
* Significant cardiopulmonary or hepatic dysfunction
* Hypersensitivity to study medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Norton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine | Esmolol | Placebo
Started | 13 | 13 | 7
Completed | 11 | 10 | 6
Not Completed | 2 | 3 | 1
Not completed — PIV in location that was excluded, surgery cancelled | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Esmolol | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 7 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.21) | 44.9 (14.05) | 48.57 (10.76) | 47.39 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: PIV in location that was excluded, surgery cancelled
  BMI exclusion, surg cx, exclusionary med to be used
  exclusionary med to be used
  Participants
    number analyzed (Participants) | 11 | 10 | 6 | 27
    Female | 9 | 5 | 3 | 17
    Male | 2 | 5 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: PIV in location that was excluded, surgery cancelled
  BMI exclusion, surg cx, exclusionary med to be used
  exclusionary med to be used
  Participants
    number analyzed (Participants) | 11 | 10 | 6 | 27
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 1 | 3 | 0 | 4
    White | 10 | 0 | 5 | 15
    More than one race | 0 | 5 | 0 | 5
    Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Score
Description: pain scoring system previously used by studies looking at various remedies to decrease Propofol injection pain - 0-10 with 0=no pain up to 10=worst pain imaginable
Time Frame: following administration of a sub-induction dose of propofol, 0.5 mg/kg up to 50 mg, just prior to full induction
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine | Esmolol | Placebo
Number analyzed (Participants) | 11 | 10 | 6
score on a scale | 0.45 (0.66) | 0.5 (1.02) | 1.83 (1.07)

2. Secondary Outcome: Heart Rate
Description: heart rate is measured as numbers on a scale with normal 60-100
Time Frame: heart rate is measured each minute for the first 10 minutes following induction
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Lidocaine | Esmolol | Placebo
Number analyzed (Participants) | 11 | 10 | 6
beats per minute
  Minute 2 | 72.6 (12.2) | 81 (14.25) | 82 (11.15)
  Minute 3 | 72.4 (14.18) | 82 (17.46) | 77.2 (11.33)
  Minute 4 | 76.9 (13.37) | 78.4 (13.14) | 79 (11.5)
  Minute 5 | 76.8 (16.99) | 91.7 (26.54) | 83.3 (10.89)
  Minute 6 | 77.4 (15.62) | 84 (10.92) | 86 (10.13)
  Minute 7 | 83.3 (24.25) | 89.5 (12.41) | 84.3 (11.76)
  Minute 8 | 75.5 (13.43) | 83.4 (13.8) | 80.5 (10.75)
  Minute 9 | 73.6 (15.46) | 85.2 (8.98) | 80.8 (8.3)
  Minute 10 | 72.18 (17.02) | 80.2 (12.59) | 83.7 (21.05)

3. Secondary Outcome: Systolic Blood Pressure
Description: blood pressure measured in mmHg
Time Frame: Systolic Blood Pressure is measured each minute for the first 10 minutes following induction
Measure: Mean (Standard Deviation); unit: mm Hg (millimeters of mercury)
Arm/Group | Lidocaine | Esmolol | Placebo
Number analyzed (Participants) | 11 | 10 | 6
mm Hg (millimeters of mercury)
  Minute 2 | 122.7 (18.15) | 126 (26.45) | 147.2 (33.45)
  Minute 3 | 116.1 (22.77) | 114 (23.6) | 153.3 (31.78)
  Minute 4 | 121.6 (12.19) | 112 (20.52) | 134.4 (17.94)
  Minute 5 | 115.4 (14.45) | 110.5 (18.59) | 123.8 (21.47)
  Minute 6 | 117.9 (10.31) | 138.6 (29.79) | 136.5 (52.49)
  Minute 7 | 121.2 (20.79) | 140.9 (37.29) | 128.8 (37.33)
  Minute 8 | 113.8 (15.52) | 127.1 (27.54) | 137 (43.08)
  Minute 9 | 116.8 (6.94) | 122.4 (26.09) | 126 (29.81)
  Minute 10 | 108 (12.17) | 117 (18.42) | 128.4 (30.88)

4. Secondary Outcome: Oxygen Saturation Percentage
Description: oxygen saturation is measured on a percentage, with normal range >90%
Time Frame: Oxygen saturation measured each minute for the first 10 minutes following induction
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Lidocaine | Esmolol | Placebo
Number analyzed (Participants) | 11 | 10 | 6
percentage
  Minute 2 | 99.6 (0.64) | 99.9 (0.3) | 99.8 (0.37)
  Minute 3 | 99.6 (0.64) | 99.89 (0.31) | 99.8 (0.37)
  Minute 4 | 99.5 (0.66) | 99.9 (0.3) | 99.8 (0.37)
  Minute 5 | 99.2 (1.19) | 99.9 (0.3) | 99.8 (0.37)
  Minute 6 | 99.2 (1.19) | 99.89 (0.31) | 99.2 (0.9)
  Minute 7 | 99.2 (1.19) | 99.7 (0.46) | 99.3 (0.47)
  Minute 8 | 98.8 (1.47) | 99.6 (0.66) | 99 (1.16)
  Minute 9 | 99.2 (1.19) | 99.9 (0.31) | 99.5 (0.76)
  Minute 10 | 99.3 (1.14) | 99.7 (0.64) | 99.3 (0.94)

ADVERSE EVENTS:
Time Frame: 10 minutes
Arm/Group | Lidocaine | Esmolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04356352/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04356352/ICF_000.pdf